CLINICAL TRIAL: NCT01074398
Title: ERCC1 Expression as a Predictor of Progression Free and Overall Survival in Patients With Epithelial Ovarian Cancer Treated on GOG Protocols 0172 and 0182
Brief Title: Biomarkers in Predicting Response in Patients With Advanced Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer Treated on GOG-0172 or GOG-0182
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Philip J. DiSaia, Gynecologic Oncology Group
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000663840; GOG-8012
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis; Immunohistochemistry

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: polymorphism analysis
Genetic: protein expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is looking at biomarkers in predicting response in patients with advanced ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate ERCC1 tumor expression, as measured by IHC, as a predictor of progression-free and overall survival of patients with advanced ovarian epithelial cancer.

Secondary

* To correlate ERCC1 single-nucleotide polymorphisms (C8092A and codon 118) with ERCC1 tumor expression.

OUTLINE: This is a multicenter study.

Blood and paraffin-embedded tumor tissue samples are analyzed for ERCC1 tumor expression by IHC and single-nucleotide polymorphisms.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced invasive ovarian epithelial carcinoma, fallopian tube adenocarcinoma, or primary peritoneal carcinoma
* Has undergone optimal surgical staging
* Has received chemotherapy on either GOG-0172 or GOG-0182
* Adequate blood or DNA available for ERCC1 analysis
* Adequate tumor on paraffin-embedded tissue for IHC staining

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Association between ERCC1 tumor expression and progression-free and overall survival

SECONDARY OUTCOMES:
Association between ERCC1 polymorphisms and ERCC1 tumor expression

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Krivak, MD, Study Chair — University of Pittsburgh

REFERENCES:
- [Derived] Rose PG, Java JJ, Salani R, Geller MA, Secord AA, Tewari KS, Bender DP, Mutch DG, Friedlander ML, Van Le L, Method MW, Hamilton CA, Lee RB, Wenham RM, Guntupalli SR, Markman M, Muggia FM, Armstrong DK, Bookman MA, Burger RA, Copeland LJ. Nomogram for Predicting Individual Survival After Recurrence of Advanced-Stage, High-Grade Ovarian Carcinoma. Obstet Gynecol. 2019 Feb;133(2):245-254. doi: 10.1097/AOG.0000000000003086. PMID 30633128